CLINICAL TRIAL: NCT04062877
Title: Clinical Transformation Application and Technology Research in Liquid Biopsy for Precise Diagnosis and Prognosis of Lymphoma
Brief Title: Clinical Application of Liquid Biopsy for Precise Diagnosis and Prognosis in Lymphoma
Status: Completed | Type: Observational
Sponsor: Ge Zheng (Other)
Responsible Party: Sponsor-Investigator, Ge Zheng, Director of Department of Hematology, Zhongda Hospital
Organization: Zhongda Hospital (Other)
Other Study IDs: ZDYYGZ201907
Record Dates: First submitted 2019-08-05; First posted 2019-08-20 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Lymphoma
Keywords: Fluid biopsy; lymphoma; accurate diagnosis
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — patients'samples from peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lymphoma is a highly heterogeneous blood malignancy. It is very important to search for relative specific diagnostic markers that can detect related lymphoma in early stage for the treatment and long-term prognosis of the disease, as the hematopoietic diseases, such as lymphoma, are more difficult to biopsy than solid tumors, with more damage and side effects.Liquid Biopsy (Liquid Biopsy) refers to the extraction of solid biological tissue, is the most common blood, also including saliva, urine, cerebrospinal fluid and other body fluids, and extract the circulating tumor cells (circulating tumor cell, CTC) and circulating tumor DNA (circulating tumor DNA, ctDNA) is used to assess related diseases. CTCs/CSCs have the ability to generate new tumors and play a key role in tumor metastasis.This project intends to develop liquid biopsy technology for accurate diagnosis and prognosis judgment of lymphoma, to carry out clinical transformation application and serve patients.

DETAILED DESCRIPTION:
1. Patients with series and matched lymphoma who were refractory to initial diagnosis, remission and recurrence were enrolled, our research group will collected patient information comprehensively and signed the informed consent.
2. The standard diagnosis process and treatment selection will be completed, and our research group willcollect relevant clinical and laboratory data.
3. 5 ml of peripheral blood from each patient was collected with EDTA anticoagulant tube, and the blood cells were centrifuged at 820×g for 10 min at 4℃ within 1 h to separate the blood cells.The plasma was then transferred to a microcentrifuge tube and centrifuged at 4℃ at 20,000×g for 10 min to remove cell debris.According to the reagent instructions, cfDNA was extracted from 2 ml cell-free plasma and the concentration of cfDNA in each patient was determined.Meanwhile, genomic DNA kit was used to extract matching tumor DNA from lymphoma bone marrow tissue.
4. We will extract the lymphoma of bone marrow tissue samples of RNA, and reverse transcription for cDNA, the use of qRT PCR verifying the mutations in tissue samples, after identifying the lymphoma five of the most common mutations from the cancer genome map (TCGA;http://cancergenome.nih.gov/) .
5. The differences of mutations detected by liquid biopsy and tumor in situ biopsy will be compared, by NGS sequencing of peripheral blood cfDNA and lymphoma tissue DNA. Meanwhile, the mutation rate of each gene mutation was analyzed for lymphoma tissue type.
6. The classification and malignant changes of matched lymphomas were statistically analyzed to study the differences in cfDNA concentration of different types of lymphomas, according to the cfDNA concentration determined at the earlier stage.
7. The mutation differences of cfDNA in the peripheral blood of each patient will be compared at three time points before, during and after treatment, combined with PET/CT detection, and the correlation between cfDNA detection indexes and therapeutic effect and prognosis monitoring will be evaluated.
8. SPSS 23.0 statistical software would be used to evaluate the correlation between cfDNA concentration in lymphoma and disease staging, grouping, subtype, efficacy prediction and recurrence monitoring. P<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* patients of lymphoma diagnosed of de novo, CR, relapsed/refractory, be willing to receive treatment

Exclusion Criteria:

* leukemia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients of lymphoma diagnosed of de novo, CR, relapsed/refractory, be willing to receive treatment, aged between 14 to 75 years.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
complete remission | From date of randomization or initial treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 weeks
  Patients achieve complete remission after initial treatment
relapse | From date of randomization or complete remission until the date of first documented relapse from any cause，assessed up to 100weeks.
  Patients' disease progress after complete remission

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Ge, Study Director — Director of Department of Hematology Zhongda Hospital
Locations (1):
- Institute of Hematology Southeast University Department of Hematology Zhongda Hospital Southeast University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided